CLINICAL TRIAL: NCT06579183
Title: A Pilot Randomized, Double-blinded, Placebo-controlled Trial on the Effects and Safety of Health Products Combining Traditional Chinese Medicines, Vitamins and Amino Acids in Psychological Distress and Insomnia
Brief Title: Pilot Trial for Health Products in Psychological Distress and Insomnia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Zhang Zhang-Jin, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 24-183
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Psychological Distress; Insomnia
Keywords: Psychological distress; Insomnia; Chinese medicine; Health product; Extra Strength VitaJoy; Extra Strength Vita Calm
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ES/VJ+ES/VC (Experimental): Participants will be instructed to orally take ES/VJ and ES/VC capsules each day, and will continue their current medications as usual, including prescribed sleep pills, anxiolytics, and antidepressants, for 12 weeks.
  Interventions: Dietary Supplement: Extra Strength VitaJoy (ES/VJ); Dietary Supplement: Extra Strength Vita Calm (ES/VC)
- Placebo (Placebo Comparator): Participants will be instructed to orally take placebo capsules each day, and will continue their current medications as usual, including prescribed sleep pills, anxiolytics, and antidepressants, for 12 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Extra Strength VitaJoy (ES/VJ) — Extra Strength VitaJoy Capsule, 2 capsules in the morning
  Arms: ES/VJ+ES/VC
Dietary Supplement: Extra Strength Vita Calm (ES/VC) — Extra Strength Vita Calm Capsule, 2 capsules in the evening
  Arms: ES/VJ+ES/VC
Dietary Supplement: Placebo — Placebo Capsule, 4 capsules in the morning and evening respectively
  Arms: Placebo

SUMMARY:
This is a pilot, single-site, two-armed, 16 weeks, double-blinded, randomized, placebo-controlled trial. A total of 60 patients aged 18-65 with psychological distress will be recruited. They will be randomly assigned to receive a combination of ES/VJ and ES/VC, or placebos (30 each) for 12 weeks. A 4-week observational phase will follow, and a post-intervention visit will be held at week 16. Written informed consent forms are obtained prior to commencement of the study from each participant. The primary outcome will be assessed using the Chinese version of the Beck Anxiety Inventory (BAI-C). The secondary outcomes include the Chinese version of the Beck Depression Inventory II (C-BDI-II) for depression, the Zung Self-Rating Anxiety Scale (SAS) as an additional assessment that measures intensity of anxiety, the Zung Self-Rating Depression Scale (SDS) as an additional assessment that measures intensity of depression, the Pittsburgh Sleep Quality Index (PSQI) for sleep quality, and the World Health Organization Quality of Life-Brief (WHOQOL-BREF) (HK version) for the general quality of life. Safety profile of ES/VJ and ES/VC will also be evaluated. A generalized linear mixed-effect model will be applied to compare outcomes over time in the 2 groups.

DETAILED DESCRIPTION:
Psychological distress is a state of emotional suffering characterized by a combination of undifferentiated symptoms ranging from anxiety (e.g., restlessness), depression (e.g., loss of interest), stress, to functional impairment. Among these symptoms, anxiety and depression, which can be subclinical symptoms or clinical diagnoses, are highly comorbid. Somatic symptoms such as insomnia, lack of energy, and headache often accompany psychological distress, too.

Psychological distress can be a precursor and/ or feature of various mental disorders, where an individual's cognition, emotional regulation, or behavior is significantly disturbed. It is highly prevalent in the general population and has become more severe during and after the COVID-19 pandemic. The global prevalence of psychological distress with insomnia has dramatically risen since the COVID-19 pandemic, with 25.6% for anxiety, 23.1% for depression, and 17.4% for insomnia. In Hong Kong, 19% suffer from depression and 14% have anxiety. However, psychological distress and insomnia are often underdiagnosed and vastly undertreated because the condition of most individuals is mild, and some fear drugs would elicit undesirable side effects, which can sometimes be a greater risk than the disease itself. The development of novel alternative treatment strategies is therefore greatly desired.

The use of Chinese medicine and complementary medicine has gained increased attention in treating mental-related disorders in recent decades. A vast number of studies have suggested the benefits of Chinese medicines, vitamins, and amino acid supplementary products in improving anxiety, depression, and insomnia. It is possible that Chinese medicines, vitamins, and amino acids together can bring about beneficial synergistic effects in treating psychological distress and insomnia.

Extra Strength VitaJoy (ES/VJ) and Extra Strength Vita Calm (ES/VC) are two health products that are formulated by combining Chinese medicines, multiple vitamins and amino acids. Chinese medicines of ES/VJ and ES/VC are developed based on traditional Chinese medicine theory, aligning with compatibility of traditional Chinese Medicine and following the basic Chinese medicine formula structure of "Jun-Chen-Zuo-Shi". The two products are thought to tranquilize anxiety and nervousness, relieve sadness and depression, and improve sleeplessness. Our preliminary animal studies have suggested that Chinese medicines of ES/VJ noticeably reduced depression-like behavior in animal models, probably via the modulation of monoamine oxidase (MAO), without inducing herb-drug interaction or hypertension. Chinese medicines of ES/VC rapidly induced sleep in animals and reduced anxiety, and their efficacy was comparable to that of benzodiazepines. A pilot clinical observation revealed that Chinese medicine preparation of ES/VC could improve multiple sleep variables recorded by Actiwatch and diary. Although determination of synergistic effects between Chinese medicine, vitamins and amino acids is not addressed in this study due to time and resource limitations, results of our preliminary studies have encouraged us to further conduct a randomized controlled trial to confirm the effects and safety of the two products, in particular anxiety and depressive symptoms and insomnia alleviation.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for this study if they:

1. are experiencing anxiety and/or depressive symptoms, as evidenced by a BAI-C score of at least 8 (no symptoms = 0-7; mild = 8-15; moderate = 16-25; severe = 26-63) and/or a C-BDI-II score of at least 14 (no symptoms = 0-13, mild = 14-19; moderate = 20-28; severe = 29-63), with symptoms persistent for more than 3 months; and
2. are able to provide informed consent for participation, take medications and complete questionnaires as scheduled.

Exclusion Criteria:

Subjects will be excluded if they:

1. have unstable systemic medical conditions that may limit their participation in the study (e.g., severe liver, cardiovascular or kidney impairment; gastrointestinal or endocrine dysfunction; malignancy; autoimmune disease or acute infectious disease);
2. have bipolar disorder, psychotic disorder (e.g., schizophrenia), organic mental disorder (e.g., Alzheimer's disease), or significant cognitive impairment;
3. present suicidal ideation (a score of ≥3 for all questionnaires of the Columbia-Suicide Severity Rating Scale (C-SSRS);
4. have a history of brain injury or surgery;
5. have alcohol abuse or substance abuse;
6. are pregnant or in lactation, or are intend to conceive;
7. have use of herbal remedies in the previous 6 months;
8. have a history of hypersensitivity to investigational drug treatment or the active or inactive constituents of the tested products;
9. have treatment with brain stimulation in the previous 6 months; or
10. are involved in other interventional clinical studies in the last 3 months or any relevant condition potentially interfering with study evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in the Beck Anxiety Inventory score | Baseline, Week 4, Week 8, Week 12, Week 16
  Beck Anxiety Inventory (BAI-C) is used to measure the severity of anxiety and its overall score ranges from 0 to 63. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8, week 12 and week 16 (post-intervention visit).

SECONDARY OUTCOMES:
Change in the Beck Depression Inventory-II score | Baseline, Week 4, Week 8, Week 12, Week 16
  Beck Depression Inventory-II (C-BDI-II) is used to measure the severity of depression and its overall score ranges from 0 to 63. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8, week 12 and week 16 (post-intervention visit).
Change in the Zung Self-Rating Anxiety Scale score | Baseline, Week 4, Week 8, Week 12, Week 16
  Zung Self-Rating Anxiety Scale (SAS) is used to measure the severity of anxiety and its overall score ranges from 25 to 100. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8, week 12 and week 16 (post-intervention visit).
Change in the Zung Self-Rating Depression Scale score | Baseline, Week 4, Week 8, Week 12, Week 16
  Zung Self-Rating Depression Scale (SDS) is used to measure the severity of depression and its overall score ranges from 25 to 100. A higher score indicates greater severity. Assessments will be conducted at baseline, week 4, week 8, week 12 and week 16 (post-intervention visit).
Change in the Pittsburgh Sleep Quality Index score | Baseline, Week 4, Week 8, Week 12, Week 16
  Pittsburgh Sleep Quality Index (PSQI) is used to assess sleep quality and its overall score ranges from 0 to 21. A higher score indicates more acute sleep disturbances. Assessments will be conducted at baseline, week 4, week 8, week 12 and week 16 (post-intervention visit).
Change in the World Health Organization Quality of Life-Brief (HK version) score | Baseline, Week 4, Week 8, Week 12, Week 16
  World Health Organization Quality of Life-Brief (WHOQOL-BREF) (HK version) is used to assess quality of life, with four quality of life domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items). Each individual item is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. A higher score indicates better quality of life. Assessments will be conducted at baseline, week 6 and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang-Jin Zhang, MMed, PhD, Principal Investigator — School of Chinese Medicine, The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Morin CM, Bjorvatn B, Chung F, Holzinger B, Partinen M, Penzel T, Ivers H, Wing YK, Chan NY, Merikanto I, Mota-Rolim S, Macedo T, De Gennaro L, Leger D, Dauvilliers Y, Plazzi G, Nadorff MR, Bolstad CJ, Sieminski M, Benedict C, Cedernaes J, Inoue Y, Han F, Espie CA. Insomnia, anxiety, and depression during the COVID-19 pandemic: an international collaborative study. Sleep Med. 2021 Nov;87:38-45. doi: 10.1016/j.sleep.2021.07.035. Epub 2021 Aug 4. PMID 34508986
- [Background] Choi EPH, Hui BPH, Wan EYF. Depression and Anxiety in Hong Kong during COVID-19. Int J Environ Res Public Health. 2020 May 25;17(10):3740. doi: 10.3390/ijerph17103740. PMID 32466251
- [Background] Sarris J, Ravindran A, Yatham LN, Marx W, Rucklidge JJ, McIntyre RS, Akhondzadeh S, Benedetti F, Caneo C, Cramer H, Cribb L, de Manincor M, Dean O, Deslandes AC, Freeman MP, Gangadhar B, Harvey BH, Kasper S, Lake J, Lopresti A, Lu L, Metri NJ, Mischoulon D, Ng CH, Nishi D, Rahimi R, Seedat S, Sinclair J, Su KP, Zhang ZJ, Berk M. Clinician guidelines for the treatment of psychiatric disorders with nutraceuticals and phytoceuticals: The World Federation of Societies of Biological Psychiatry (WFSBP) and Canadian Network for Mood and Anxiety Treatments (CANMAT) Taskforce. World J Biol Psychiatry. 2022 Jul;23(6):424-455. doi: 10.1080/15622975.2021.2013041. Epub 2022 Mar 21. PMID 35311615
- [Background] Sarris J, Marx W, Ashton MM, Ng CH, Galvao-Coelho N, Ayati Z, Zhang ZJ, Kasper S, Ravindran A, Harvey BH, Lopresti A, Mischoulon D, Amsterdam J, Yatham LN, Berk M. Plant-based Medicines (Phytoceuticals) in the Treatment of Psychiatric Disorders: A Meta-review of Meta-analyses of Randomized Controlled Trials: Les medicaments a base de plantes (phytoceutiques) dans le traitement des troubles psychiatriques: une meta-revue des meta-analyses d'essais randomises controles. Can J Psychiatry. 2021 Oct;66(10):849-862. doi: 10.1177/0706743720979917. Epub 2021 Feb 18. PMID 33596697